CLINICAL TRIAL: NCT07057986
Title: Trans-Cervical and Trans-abdominal Ultrasound for Monitoring Esophageal Thickness in Eosinophilic Esophagitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-25-2153-AL-CTIL
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Eosinophilic Esophagitis (EoE)
Keywords: eosinophilic esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with suspected or confirmed diagnosis of Eosinophilic esophagitis (Experimental): Patients will undergo trans-cervical or abdominal ultrasound before their scheduled upper endoscopy with biopsies.
  Interventions: Device: Trans cervical or abdominal ultrasound

INTERVENTIONS:
Device: Trans cervical or abdominal ultrasound — ultrasound assessment before the scheduled upper endoscopy.

SUMMARY:
Eosinophilic Esophagitis (EoE) is a chronic inflammatory disease characterized by eosinophilic infiltration of the esophageal mucosa, leading to symptoms of dysphagia and food impaction. Currently, upper endoscopy with biopsy is the gold standard for diagnosis and disease monitoring, but it is invasive, costly, and associated with procedural risks. The investigators want to use ultrasound imaging as a non-invasive assessment of esophageal wall thickness as a surrogate marker for mucosal inflammation.

Participants will undergo ultrasound assessment at the same day of endoscopy, and than after 3-6 months (optional). The correlation between US-measured esophageal thickness and histological eosinophil counts will be measured.

DETAILED DESCRIPTION:
Eosinophilic Esophagitis (EoE) is a chronic inflammatory disease characterized by eosinophilic infiltration of the esophageal mucosa, leading to symptoms of dysphagia and food impaction. Currently, upper endoscopy with biopsy is the gold standard for diagnosis and disease monitoring, but it is invasive, costly, and associated with procedural risks.

Recent advances in ultrasound (US) imaging suggest the potential for non-invasive assessment of esophageal wall thickness as a surrogate marker for mucosal inflammation. This study aims to evaluate the efficacy and accuracy of trans-cervical/abdominal ultrasound in assessing esophageal thickness compared to the conventional endoscopic evaluation in patients with suspected or confirmed EoE. If validated, this approach could significantly reduce patient burden and reliance on frequent invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Suspected or confirmed diagnosis of EoE based on clinical symptoms (e.g., dysphagia, food impaction).
* Scheduled for upper endoscopy with biopsies.
* Able and willing to consent to participation.

Exclusion Criteria:

* Prior esophageal surgery or anatomical abnormalities.
* Presence of other gastrointestinal disorders affecting the esophagus (e.g., esophageal cancer, achalasia, Barrett's esophagus).
* Pregnancy.
* Inability to undergo US due to anatomical or physical limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between US-measured esophageal thickness and Eosinophilic Esophagitis Endoscopic Reference Score / histological eosinophil counts. | 6 months
  Comparison of ultrasound results and histological results of eosinophils. Esophagitis Endoscopic Reference score scale: Fixed rings: 0-3, Exudates: 0-2, Furrows: 0-2, Oedema: 0-2, Stricture: 0-1, Feline esophagus: 0-1, Narrow calibre esophagus: 0-1, Crepe paper esophagus: 0-1. Higher scores mean a worse outcome.

IPD SHARING:
Plan to Share IPD: Yes
General baseline data Endoscopy data
Supporting Information: Study Protocol
Time Frame: Will be available at study conclusion
Access Criteria: Access by request to the PI